CLINICAL TRIAL: NCT03294863
Title: Use of Embrace Device After Cutaneous Wound Closure: a Randomized Evaluator Blinded Split Wound Comparative Effectiveness Trial
Brief Title: Effectiveness of Embrace Scar Therapy Device After Cutaneous Wound Closure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: 101077
Record Dates: First submitted 2017-09-22; First posted 2017-09-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Linear Cutaneous Wound
Keywords: Scar; Cosmesis; Embrace Device; Split Wound; Wound Closure; Cutaneous Wound
MeSH Terms: conditions — Cicatrix | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Each subject receives both types of interventions upon the same scar in order for comparison.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Embrace Scar Therapy Device (Experimental): 16x5-cm silicone elastomeric dressing that adheres to the skin using a pressure-sensitive silicone adhesive will be applied to 1/2 of the cutaneous wound
  Interventions: Device: Embrace Scar Therapy Device
- Standard of Care (Placebo Comparator): Another 1/2 of cutaneous wound will be treated per standard of care
  Interventions: Other: Standard of Care

INTERVENTIONS:
Device: Embrace Scar Therapy Device — 16x5-cm silicone elastomeric dressing that adheres to the skin using a pressure-sensitive silicone adhesive.
  Arms: Embrace Scar Therapy Device
Other: Standard of Care — Without the embrace Scar Therapy Device
  Arms: Standard of Care

SUMMARY:
The purpose of this study is to determine whether the use of the embrace device after repair of linear cutaneous surgery wounds improves scar cosmesis.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether the use of the embrace device after repair of linear cutaneous surgery wounds improves scar cosmesis. We will use a split wound model, half of the wound is treated with the embrace device and the other half is not treated. Three-months post-surgery, the scar will be measured via the physician observer scar assessment scale, a validated scar instrument. The scar width and adverse events will also be recorded.

Following the surgical repair of cutaneous wounds, scar formation is inevitable and results in varying degrees of aesthetic and/or functional impairment. Numerous treatment modalities have been employed to treat scars. Carbon dioxide and pulse dye lasers, as well as dermabrasion can reduce erythema and irregular topology of the scar surface1,2. Silicone-based products have also been used to treat post-surgical scars, including gels, sheets, and tape3-5. Intralesional steroids are often injected into to induce flattening of a scar6. More recent research has highlighted the impact of mechanical forces and tension on scar formation. In one report, incisions in both pigs and humans were treated with a tension-shielding device and showed a reduction in scarring7. More recently two clinical trials have been published in the plastic surgery literature showing that the use of the embrace device, a silicone-based dressing designed to minimize wound tension, is effective in improving the aesthetic outcome following scar revision surgery8,9. While these initial studies of the embrace device have promising findings, there are significant drawbacks to both studies including small study population, inclusion of patients seeking scar revision (a select group likely predisposed to poor scar cosmesis and not representative of first-time surgical patients), investigator conflict of interest, and the use of a digital software-based scar assessment tool using patients photos that were not standardized with respect to lighting or distance. Therefore, larger studies in first-time surgical patients with standardized photos for scar assessment are required to validate this potentially promising device for improved scar cosmesis.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Able to give informed consent themselves
* Patient scheduled for cutaneous surgical procedure along a flat surface suitable to application of the embrace with predicted primary closure.
* Able to apply dressings themselves.
* Willing to return for follow up visits.

Exclusion Criteria:

* Mentally handicapped
* Unable to understand written and oral English
* Incarceration
* Under 18 years of age
* Pregnant Women
* Wounds with predicted closure length less than 3 cm
* Patients with known adverse reactions to adhesives
* Patients with history of collagen vascular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2025-12-08 (Actual)

PRIMARY OUTCOMES:
Physician observer scar assessment score (POSAS) | 3 months
  Comparison of scar cosmesis over area of wound that was treated with the device as compared to area that was not treated with the device.
Width of the scar | 3 months
  The width of the scar on both sides will also be measured and recorded 1 cm from midline on both sides of the scar

CONTACTS AND LOCATIONS:
Overall Officials: Daniel B Eisen, MD, Principal Investigator — UC Davis
Locations (1):
- University of California, Davis, Department of Dermatology, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: Undecided